CLINICAL TRIAL: NCT04828356
Title: Assistant Professor
Brief Title: The Effect of Foot Reflexology on Pain, Comfort and Beta Endorphin Levels in Patients With Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gurkan Kapikiran, Assistant Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018/183
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Liver Transplant; Complications
Keywords: Liver Transplantation; Foot Reflexology; Pain; Comfort; Beta Endorphin
MeSH Terms: conditions — Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot reflexology group (Experimental): The first researcher received hands-on training about reflexology application before the study started. The researcher applied foot reflexology on the patients with liver transplantation in the experimental group in one session (30 minutes) after the operation. Patient confidentiality was maintained in all procedures. The patient identity form was implemented before reflexology application. Pain and comfort levels were assessed as the pre-test. Then, venous blood was taken to determine the plasma β-End level. Foot reflexology was first applied on the right foot, which is effective on the sympathetic nervous system, for 15 min and then, on the left foot, which is effective on the parasympathetic nervous system, for 15 min. Same process was performed on the left foot and the reflexology application was completed within 15 min. Venous blood was taken again to assess the β-End level as the post-test after the application, and the NPS and PCQ were implemented again.
  Interventions: Other: Reflexology
- No treatment group (No Intervention): The patient identity form, NPS and PCQ were applied on the patients in the control group as the pre-test. After the questions were answered, venous blood was taken to determine the plasma β-End level. No intervention other than clinical protocol was applied on the control group, and after taking venous blood after 30 minutes to determine β-End level, the NPS and PCQ were re-applied as the post-test.

INTERVENTIONS:
Other: Reflexology — Reflexology application is an energy balancing system with its own pressure technique that provides recovery by rubbing the reflex (nerve endings) points, stroking and applying pressure during squeezing movements. Thanks to the pressure and massage applied to the reflex points, the energy blockages are broken and this energy flow is distributed in a balanced way to the relevant organs.
  Arms: Foot reflexology group

SUMMARY:
Reflexology application is an effective method in pain control by stimulating the release of endorphins. The Research was carried out to determine the effect of foot reflexology applied to patients with liver transplantation on pain, comfort and beta endorphin levels.The research was carried out as a randomized controlled study. The population of the study was made up of adult patients who underwent liver transplantation a Liver Transplant Institute in Turkey. The sample consisted of 120 patients with specified power analysis, including analysis 60 experimental and 60 controls. Data were collected between October 2019-April 2020 using Patient Information Form, Numerical Pain Scale, Perianesthesia Comfort Scale and Beta Endorphin Level Registration Form.

DETAILED DESCRIPTION:
This study was conducted in an randomized control trial, pre-test/post-test control group design. The study was conducted in an organ transplantation clinic of the Liver Transplantation Institute (LTI) in Turkey between December 2018 and July 2020. Approximately 225 liver transplantations are performed in the LTI in a year.

The population of the study included 147 patients who received liver transplantations in the LTI. The sample size was determined with the G Power 3.1.9.7 program. According to the performed power analysis measurement with 0.7 effect size, 0.05 margin of error, 0.95 confidence interval and 95% power to represent the universe, it was determined that 120 patients (60 in the experimental group, 60 in the control group) should be included in the study. The research protocol was designed according to the CONSORT (Consolidated Standards of Reporting Trials Statement) guidelines. The sample included the patients who met the inclusion criteria and who were selected from the population with the improbable random sampling method. 16 patients who did not meet the inclusion criteria and 11 patients who did not agree to participate in the study were excluded from the study.

Numbers from 1 to 120 were randomly divided into two blocks according to the algorithm created by the computer program. The blocks for the experimental and control groups were determined by lottery method. The first block was determined to be the control group while the second block was determined to be the experimental group.

Inclusion criteria were being: (i) 18 years of age or older, (ii) ability to communicate verbally and not having a cognitive problem, (iii) defining pain severity of 4 and above, and (iv) willing to participate in the study. The exclusion criteria were having: (i) the absence of open wounds and cellulite in the area to be applied, (ii) the absence of thrombophlebitis, deep vein thrombosis, inflammatory diseases, etc., and (iii) psychiatric illness.

Experimental Group The first researcher received hands-on training about reflexology application before the study started. The researcher applied foot reflexology on the patients with liver transplantation in the experimental group in one session (30 minutes) after the operation. Patient confidentiality was maintained in all procedures. It was ensured that the environment was as quiet and calm as possible for the concentration of the researcher and the patient during the application. Television and monitor sounds were reduced and phone tones were muted and turned to silent mode. The patient was asked to lie down in supine position and the researcher prepared the patient for reflexology by supporting their feet with a pillow. After completing all preparations and washing her/his hands, the researcher took some petroleum jelly and rubbed her/his hands and brought it to body temperature. The patient identity form was implemented before reflexology application. Pain and comfort levels were assessed as the pre-test. Then, venous blood was taken to determine the plasma β-End level. Foot reflexology was first applied on the right foot, which is effective on the sympathetic nervous system, for 15 min and then, on the left foot, which is effective on the parasympathetic nervous system, for 15 min. Foot warm-up movements, which are the first step of foot reflexology, were applied on the right foot for 2 min. Then, the warm-up movements were ended by applying deep and painless pressure on the solar plexus area of the foot, on which reflexology was applied, for 1 min. Then, reflexology was applied on brain (epiphysis area on the the thumb, hypothalamus, pituitary points), liver, thyroid, small and large bowels, knee, hip, elbow and shoulder areas and lymphatic system areas. Relaxation movements were then performed, and the session on the right foot session was completed within 15 minutes with the application of pressure on the solar plexus. Same process was performed on the left foot and the reflexology application was completed within 15 min. Venous blood was taken again to assess the β-End level as the post-test after the application, and the NPS and PCQ were implemented again.

Control (No treatment) Group The patient identity form, NPS and PCQ were applied on the patients in the control group as the pre-test. After the questions were answered, venous blood was taken to determine the plasma β-End level. No intervention other than clinical protocol was applied on the control group, and after taking venous blood after 30 minutes to determine β-End level, the NPS and PCQ were re-applied as the post-test.

Laboratory Analyses Venous blood was taken from the patients on the 0 and 30 minutes to measure the β-End level. 5 mL venous blood sample taken from each patient with a sterile single-use 10 cc injector was poured into gold BD Hemogard capped tubes. Blood samples were kept upright at room temperature for 15-20 minutes, then they were centrifuged at +4 ° C, 2000-3000 gauge for 20 minutes. Following the centrifugation, the separated serum was taken from the tubes and stored in Eppendorf tubes at -80 ° C. After completing taking blood samples, serums were thawed and studied in accordance with the kit package insert (Catalog No: YL191012375, YL191012376, YL191012377) to determine β-End level. The laboratory analyses were performed by experts in the Microbiology Department Laboratory of a university.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Ability to communicate verbally and not having a cognitive problem
* Defining pain severity of 4 and above
* Willing to participate in the study.

Exclusion Criteria:

* The absence of open wounds and cellulite in the area to be applied
* The absence of thrombophlebitis, deep vein thrombosis, inflammatory diseases
* Psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Scale | 0.-30. minutes
  It is a numeric scale which is based on explaining pain severity with numbers, and where 0 point means no pain and 10 points mean unbearable pain
Beta-Endorphin Level Entry Form | 0.-30. minutes
  This form, in which the β-End level determined after laboratory analysis is recorded, was established by the researcher.
Perianesthesia Comfort Questionnaire (PCQ) | 0.-30. minutes
  PCQ was established based on the taxonomic structure which forms the hypothetical components of the comfort hypothesis

CONTACTS AND LOCATIONS:
Locations (1):
- Gürkan, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided